CLINICAL TRIAL: NCT01365936
Title: Influence of Ovarian Stimulation With hMG or Recombinant FSH on OHSS Prevention in PCOS Patients Undergoing IVF
Brief Title: hMG or Recombinant FSH on OHSS Prevention in PCOS Patients Undergoing IVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Figen Turkcapar, MD, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZTBIVF1
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: IVF; ICSI; OHSS; PCOS; recFSH; HMG
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- menotrophin (Active Comparator): In this prospective trial, women with PCOS (according to Rotterdam criteria) were randomized (80 patients) after GnRH analogue suppression to stimulation with HMG (n=38) or rFSH (n=42) using a low dose step up protocol in ICSI cycles.
  Interventions: Drug: HMG
- recombinant FSH (Active Comparator): Patients were randomized after GnRH analogue suppression to stimulation with HMG (n=38) or rFSH (n=42) using a low dose step up protocol in ICSI cycles.
  Interventions: Drug: rFSH

INTERVENTIONS:
Drug: HMG — In this prospective trial, women with PCOS (according to Rotterdam criteria) were randomized (80 patients) after GnRH analogue suppression to stimulation with HMG (n=38) or rFSH (n=42) using a low dose step up protocol in ICSI cycles.
  Other Names: Menotrophin
  Arms: menotrophin
Drug: rFSH — Patients were randomized after GnRH analogue suppression to stimulation with HMG (n=38) or rFSH (n=42) using a low dose step up protocol in ICSI cycles.
  Arms: recombinant FSH

SUMMARY:
There have been some controversies regarding the use of preparations with LH activity in patients with polycystic ovary syndrome (PCOS) who have high endogenous LH activity. In this research we aimed to compare urinary menotrophin versus recombinant FSH (rFSH) with respect to the prevention of OHSS

DETAILED DESCRIPTION:
Polycystic ovary syndrome was diagnosed according to the Rotterdam criteria. Patients older than 38 years or with serum FSH level ≥12mIU/ml and a history of ovarian surgery were excluded from the study. All of our patients were given combined oral contraceptive (Yasmin) prior to ovulation induction cycles. Leuprolide Acetate (Lucrin daily; Abbott, Istanbul) therapy was started in mid-luteal phase to induce pituitary down regulation, and was initiated at a dose of 1.0 mg SC daily until pituitary down-regulation was established. The leuprolide acetate dose was then reduced to 0.5 mg daily until the day of human chorionic gonadotropin (hCG) administration. After GnRH analogue suppression was achieved, the patients were randomized using block randomization (block of two) to stimulation with hMG (Menogon; Ferring Pharmaceuticals. Istanbul) or rFSH (Gonal-F; Serono Istanbul). Starting dose was 150IU for the first 3 days of stimulation, after which daily dosing was determined individually. Serial Estrodiol (E2) levels and two-dimensional follicle measurements by transvaginal ultrasonography (LOGIC 200 PRO, General Electric, Korea) were performed until at least two dominant follicles reached dimensions of 18 mm or greater in diameter. Human chorionic gonadotropin (Pregnyl, Organon, 10,000 IU- IM) was then administered, followed by transvaginal oocyte retrieval 36 hours later. The criteria of coasting in our institute were serum E2 >3600 pg/ml and multiple intermediate follicle. During coasting period, gonadotropin was withheld, but leuprolide acetate was continued at 0.5mg/d. ICSI was performed for all the patients. Fertilization was assessed at 20h (±1h), and embryo quality was assessed at 28, 44, and 68h (±1h) after oocyte retrieval. A top- quality embryo was defined as four to five cells on day 2, seven or more cells on day 3, and no multinucleation. Vaginal progesterone gel 90 mg/day 8% (Crinone;Serono) for luteal support was given from the oocyte retrieval until the clinical pregnancy (9-10 weeks of gestation) or negative serum βhCG test (13-15 days after embryo transfer).

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS

Exclusion Criteria:

* Patients older than 38 years or with serum FSH level ≥12mIU/ml and a history of ovarian surgery were excluded from the study

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
the incidence of OHSS | 6 Months
peak serum E2 levels | 6 months

SECONDARY OUTCOMES:
the need of coasting, | 6 months
number of intermediate follicles | 6 months
fertilization rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Figen A Turkcapar, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Training Hospital
Locations (1):
- Zekai Tahir Burak women's research and Training Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Figen Turkcapar A, Seckin B, Onalan G, Ozdener T, Batioglu S. Human Menopausal Gonadotropin versus Recombinant FSH in Polycystic Ovary Syndrome Patients Undergoing In Vitro Fertilization. Int J Fertil Steril. 2013 Jan;6(4):238-43. Epub 2013 Mar 3. PMID 24520446